CLINICAL TRIAL: NCT07061938
Title: Phase 1b/2a Prospective, Open Label, Multicenter, Single Arm Study to Assess Safety, Efficacy and Persistence of ACE1831, in Subjects With Immunoglobulin G4-Related Disease
Brief Title: Study to Assess Safety, Efficacy and Persistence of ACE1831, in Subjects With IgG4-Related Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acepodia Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE1831-201
Record Dates: First submitted 2025-05-27; First posted 2025-07-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: IgG4 Related Disease
Keywords: IgG4 Related Disease; cell therapy; IgG4-RD; ACE1831
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm trial (Experimental): The single, open label study arm includes 3 dose escalation cohorts:
  * Cohort 1:
    * Cohort 1a: Receives ACE1831 (Dose Level 1) with lymphodepletion conditioning (LDC)
    * Cohort 1b: Receives ACE1831 (Dose Level 1) without LDC.
  * Cohort 2: Receives ACE1831 (Dose Level 2) with or without LDC depending on assignment
  * Cohort 3: Receives ACE1831 (Dose Level 3) with or without LDC depending on assignment
  Interventions: Drug: ACE1831; Drug: Lymphodepleting chemotherapy

INTERVENTIONS:
Drug: ACE1831 — ACE1831 is allogeneic gamma delta T (gdT) cell therapy. Subjects will receive ACE1831 dose based on the assigned dose escalation cohort.
Drug: Lymphodepleting chemotherapy — Subjects assigned to receive lymphodepleting preconditioning (LDC) will receive chemotherapy cyclophosphamide ahead of ACE1831 administration.

SUMMARY:
ACE1831 is an off-the-shelf, allogeneic gamma delta T (gdT) cell therapy derived from healthy donors, that is under investigation for the treatment in subjects with Immunoglobulin G4 Related Disease (IgG4-RD)

DETAILED DESCRIPTION:
ACE1831-201 study is an Open Label, Multicenter, Single Arm Study to Assess Safety, Efficacy and Persistence of ACE1831, in Subjects with Immunoglobulin G4-Related Disease

ELIGIBILITY:
Inclusion Criteria: To be eligible for this study, all of the following inclusion criteria must be met:

* Signed Informed Consent
* Male or female ≥ 18 to 75 years of age
* Active IgG4-RD flare at screening with IgG4-RD Responder Index at least 2, confirmed by symptoms, labs, and/or imaging.
* History of IgG4-RD involving at least 2 organs/sites, and current flare involves at least 1 organ/site (excluding lymph nodes) requiring treatment.
* Elevated serum IgG4 above the upper limit of normal at screening.
* Able to receive glucocorticoids for current flare and taper to 0 mg by Day -5.
* Contraception agreement per protocol from screening through 24 weeks after last ACE1831 dose (no LDC) or 12 months after last LDC dose (with LDC).
* For sites in China only: prior treatment failure to glucocorticoids and at least one immunosuppressive agent.

Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this trial.

* Significant conditions that impair ability to receive study treatment or comply.
* Predominant fibrosis in affected organs.
* Active/latent infection that would interfere with therapy (including HBV, HCV, HIV, TB, syphilis) or significant recent infection per protocol.
* Known immunodeficiency state.
* NYHA class III/IV heart disease.
* Severe allergy/hypersensitivity to monoclonal antibodies or relevant study agents.
* Malignancy within 5 years (protocol exceptions apply).
* Recent investigational agent exposure.
* Recent B-cell depleting therapy (anti-CD20/anti-CD19) unless reconstitution per protocol.
* Live/attenuated vaccine within 2 months.
* Pregnant or breastfeeding.
* Inadequate organ function/blood counts per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of ACE1831 as Assessed by Adverse Events, Clinical Laboratory Tests, Physical Examinations, ECGs, and Vital Signs | up to 72 weeks post last-ACE1831 dose
  Primary Outcome Measures: Safety and Tolerability of ACE1831. Adverse Events: Incidence of TEAEs, SAEs, AESIs, and DLTs. Clinical Laboratory Abnormalities: Number of subjects with clinically significant abnormalities in protocol-defined clinical laboratory assessments compared with baseline.
  Physical Examination Abnormalities: Number of subjects with clinically significant changes from baseline.
  ECG Abnormalities: Number of subjects with clinically significant ECG changes (PR, QRS, QT/QTcF, heart rate) from baseline.
  Vital Signs Abnormalities: Number of subjects with clinically significant changes from baseline.
  Number of Subjects With Clinically Significant Changes in Vital Signs From Baseline. Number of subjects with clinically significant changes in vital signs, including temperature, respiratory rate, heart rate, blood pressure, and oxygen saturation (SpO₂), compared with baseline.
  For all of the above, Unit of Measure: Number of Subjects

SECONDARY OUTCOMES:
To assess the efficacy of ACE1831 (primary efficacy) | 24 weeks after last dose of ACE1831
  • Proportion of subjects in complete remission 24 weeks after last dose of ACE1831
3.1 To assess the efficacy of ACE1831 (secondary efficacy): Proportion of subjects who experience sustained complete remission | up to 72 weeks post-last ACE1831 dose
  Proportion of subjects who experience sustained complete remission 72 weeks after last dose of ACE1831
3.2 To assess the efficacy of ACE1831 (secondary efficacy): Time to first flare | up to 72 weeks post-last ACE1831 dose
  Time (days) from first dose of ACE1831 to first flare
3.3 To assess the efficacy of ACE1831 (secondary efficacy): Cumulative GC usage | up to 72 weeks post-last ACE1831 dose
  Cumulative GC usage (milligrams) at 24 weeks after the last dose of ACE1831
3.4 To assess the efficacy of ACE1831 (secondary efficacy): Changes in SF-12 | up to 72 weeks post-last ACE1831 dose
  Changes in Quality of Life Questionnaire (QOL) Short Form 12 (SF-12) total score
3.5 To assess the efficacy of ACE1831 (secondary efficacy): Changes in PGA | up to 72 weeks post-last ACE1831 dose
  Changes in Physician's Global Assessment (PGA) of disease activity score (Visual Activity Score, scale range 0 -100)
3.6 To assess the efficacy of ACE1831 (secondary efficacy): Time to PGA = 0 | up to 72 weeks post last-ACE1831 dose
  Time (days) to PGA assessment score of 0
3.7 To assess the efficacy of ACE1831 (secondary efficacy): Changes in SGA | up to 72 weeks post last-ACE1831 dose
  Changes in Subject's Global Assessment (SGA) of disease activity score (Visual Activity Score, scale range 0 - 100)
3.8 To assess the efficacy of ACE1831 (secondary efficacy): Changes in SSI | up to 72 weeks post last-ACE1831 dose
  Changes in IgG4-RD symptom severity index (IgG4-RD-SSI) score
3.9 To assess the efficacy of ACE1831 (secondary efficacy): Changes in IgG4-RD RI | up to 72 weeks post last-ACE1831 dose
  Changes in IgG4-RD Responder Index (IgG4-RD RI) score

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No